CLINICAL TRIAL: NCT07077083
Title: A Pilot Study of 89Zr-girentuximab for PET Imaging in Residual or Recurrent Post Ablative Tumors in Patients With Renal Cell Carcinoma.
Brief Title: CAIX PET/CT for Residual or Recurrent Post-ablative ccRCC
Acronym: CAIX PET/CT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Telix Pharmaceuticals, Ltd (Unknown)
Responsible Party: Principal Investigator, Shadi Abdar Esfahani, Director of Nuclear Medicine Clinical Trials, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-240
Record Dates: First submitted 2025-06-24; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Clear Cell Renal Cell Carcinoma (ccRCC); ccRCC
Keywords: kidney; kidney cancer; imaging
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patients with known or suspected recurrent or residual ccRCC (Experimental): PET and Histological correlation
  Interventions: Drug: 89Zr-Girentuximab
- Patients with ccRCC undergoing ablation (Experimental): PET for evaluation of post-ablative kidney
  Interventions: Drug: 89Zr-Girentuximab

INTERVENTIONS:
Drug: 89Zr-Girentuximab — 89Zr-Girentuximab PET

SUMMARY:
The goal of this clinical trial is to learn whether 89Zr-Girentuximab PET scans can inform management of renal cell carcinoma. The main questions it aims to answer are:

* Does the 89Zr-Girentuximab PET detect ccRCC that is left behind or has come back after treatment?
* What differences can be seen on the 89Zr-Girentuximab PET before and after standard of care treatment?

Participants in arm 1 will be given the study drug followed by a PET scan 3-7 days after injection. Participants in arm 2 will receive the same, but will proceed with their standard of care cryoablation after the initial PET scan. Within 3 days of the cryoablation treatment, participants will receive a repeat PET scan.

ELIGIBILITY:
Inclusion Criteria:

1. Written and voluntarily given Informed Consent
2. ≥18 years of age at time of consent

   a. Because no dosing or adverse event data are currently available on the use of 89Zr-girentuximab in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
3. Have the capacity to understand the study and be willing and able to comply with all protocol requirements.
4. Findings suspicious for post-ablation residual or recurrent ccRCC (subjects in cohort 1) documented at conventional imaging or biopsy, performed within 90 days prior to 89Zr-girentuximab PET scan.
5. Findings suspicious for primary ccRCC (subjects in cohort 2) documented at standard histology or conventional imaging, performed within 90 days prior to 89Zr-girentuximab PET scan.
6. Negative serum or urine pregnancy tests in female patients of childbearing potential within 72 hours prior to receiving 89Zr-girentuximab. Female patients of non-child bearing potential must provide evidence by fulfilling one of the following criteria at screening:

   1. Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   2. Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution
   3. Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy but not tubal ligation
7. For all participants, consent to practice double-barrier contraception until a minimum of 42 days after 89Zr-girentuximab administration.

Exclusion Criteria:

1. Renal mass known to be a metastasis of another primary tumor.
2. Active non-renal malignancy requiring therapy during and up to EOT visit.
3. Planned antineoplastic therapies (for the period between IV administration of 89Zr-girentuximab and imaging).
4. Previous administration of any radionuclide within 10 of its half-lives before 89Zr-girentuximab injection day.
5. Serious non-malignant disease (e.g., psychiatric, infectious, autoimmune, or metabolic), that may interfere with the objectives of the program or with the safety or compliance of the subject, as judged by the Investigator.
6. Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the program.
7. Women who are pregnant or breastfeeding.
8. Known hypersensitivity to girentuximab or DFO (desferoxamine).
9. Renal insufficiency with estimated glomerular filtration rate eGFR ≤ 40 mL/min/ 1.73 m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
SUVmean of the ablated zone and adjacent or contralateral uninvolved kidney | From enrollment to 0-3 days after SOC cryoablation
  Qualitative and quantitative assessment of 89Zr-girentuximab probe uptake of the ablative zone in the kidney will be performed. Guided by the findings of standard CT or MRI, a region of interest (ROI) will be drawn over the ablation zone and adjacent uninvolved kidney. SUVmean of the ROIs will be measured for the recurrent/residual tumor and the adjacent or contralateral normal kidney. Descriptive statistics including the mean SUVmean and standard deviation will be reported for each ROI. Tumor to kidney uptake ratio will also be calculated. It is expected that the recurrent/residual tumor will show uptake above the uninvolved kidney.
SUVmax of the ablated zone and adjacent or contralateral uninvolved kidney | From enrollment to 0-3 days after SOC cryoablation
  Qualitative and quantitative assessment of 89Zr-girentuximab probe uptake of the ablative zone in the kidney will be performed. Guided by the findings of standard CT or MRI, a region of interest (ROI) will be drawn over the ablation zone and adjacent uninvolved kidney. SUVmax of the ROIs will be measured for the recurrent/residual tumor and the adjacent or contralateral normal kidney. Descriptive statistics including the SUVmax and standard deviation will be reported for each ROI. Tumor to kidney uptake ratio will also be calculated. It is expected that the recurrent/residual tumor will show uptake above the uninvolved kidney.

SECONDARY OUTCOMES:
Comparison of SUVmean on pre- and post-ablation scans | Baseline through 0-3 days days after SOC cryoablation
  Guided by the standard CT or MRI, an ROI will be defined over the primary kidney tumor and adjacent uninvolved kidney on the scans before and after cryoablation. SUVmean as well as tumor to kidney ratio will be calculated on the pre- and post-ablation scans to evaluate whether the uptake decreases immediately after ablation.
Comparison of SUVmax on pre- and post-ablation scans | Baseline through 0-3 days after SOC cryoablation
  Guided by the standard CT or MRI, an ROI will be defined over the primary kidney tumor and adjacent uninvolved kidney on the scans before and after cryoablation. SUVmax as well as tumor to kidney ratio will be calculated on the pre- and post-ablation scans to evaluate whether the uptake decreases immediately after ablation.

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Abdar Esfahani, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The information on patient demographics, cancer (ccRCC) history, imaging findings, and histological assessment will be shared in scientific presentations and publications.